CLINICAL TRIAL: NCT07372040
Title: Clinical Study Comparing Empagliflozin, Acetazolamide, and Metolazone as Add-on Therapies to Loop Diuretics in Acute Decompensated Heart Failure
Brief Title: Add-on Diuretics in Acute Decompensated Heart Failure
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dalia Abdelhamid Gomaa, assistant lecturer of clinical pharmacy, faculty of pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acute Heart Failure 2026
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Empagliflozin; Acetazolamide; Metolazone; Acute heart failure; Add-on therapies to Loop diuretics
MeSH Terms: interventions — empagliflozin; Acetazolamide; Metolazone

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Empagliflozin group (Active Comparator): will include 22 patients who will receive 10 mg oral empagliflozin administered simultaneously with the first dose of loop diuretics each day for 3 days
  Interventions: Drug: empagliflozin
- Acetazolamide group (Active Comparator): will include 22 patients who will receive 500 mg oral acetazolamide administered simultaneously with the first dose of loop diuretics each day for 3 days
  Interventions: Drug: Acetazolamide
- Metolazone group (Active Comparator): will include 22 patients who will receive 5 mg oral metolazone administered simultaneously with the first dose of loop diuretics each day for 3 days
  Interventions: Drug: metolazone

INTERVENTIONS:
Drug: empagliflozin — Empagliflozin may augment the natriuretic and aquaretic actions of loop diuretics in patients with acute decompensated heart failure and it does not typically cause electrolyte disturbances and has been shown to improve outcomes in patients with heart failure
  Arms: Empagliflozin group
Drug: Acetazolamide — Acetazolamide can augment the action of loop diuretics in patients with acute decompensated heart failure
  Arms: Acetazolamide group
Drug: metolazone — Metolazone can augment the action of loop diuretics in patients with acute decompensated heart failure
  Arms: Metolazone group

SUMMARY:
The aim of this study is to compare the efficacy and safety of empagliflozin, acetazolamide, and metolazone as add-on therapies to loop diuretics in patients with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients older than 18 years.
2. Hospital admission with clinical diagnosis of acute decompensated heart failure with at least one clinical sign of volume overload (e.g. edema, ascites confirmed by echography or pleural effusion confirmed by chest X-ray or echography).

Exclusion Criteria:

1. Type 1 diabetes.
2. Chronic kidney disease with estimated glomerular filtration rate (eGFR) <30 mL/min per 1.73 m² or end-stage kidney failure with the need for chronic dialysis treatment.
3. A systolic blood pressure of less than 90 mmHg.
4. Cardiogenic shock.
5. Receipt of acetazolamide maintenance therapy.
6. Receipt of an SGLT2 inhibitor, thiazide, or thiazide-like diuretic in the 48 hrs before randomization.
7. Any cause of heart failure leading to decompensation that will need urgent management (eg, acute coronary syndrome, unstable arrhythmias, acute pulmonary embolism).
8. Pregnant or breastfeeding women.
9. Moderate to severe anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
The cumulative urine output measured over 3 days | 3 days

SECONDARY OUTCOMES:
- The change in serum level of N-terminal pro-brain natriuretic peptide (NT-proBNP) | 4 days
  Blood samples will be collected at baseline and after 4 days
The change in serum level of Soluble suppression of tumorigenicity 2 (sST2) | 4 days
  Blood samples will be collected at baseline and after 4 days
The change in urinary level of Tissue inhibitor of metalloproteinases-2 (TIMP-2 ) | 3 days
  Urine samples will be collected at baseline and after 3 days
The change in urinary level of Insulin-like growth factor-binding protein 7 (IGFBP7) | 3 days
  Urine samples will be collected at baseline and after 3 days
30-day mortality | up to 30 days
  Proportion of patients who die within 30 days of randomization
Proportion of patients achieving an ADVOR Score ≤ 1 without the need for escalating diuretic strategy | 3 days
  the treating physician will calculate the congestion score, on a scale from 0 to 10 on the basis of the sum of scores for the degree of edema (0 to 4), pleural effusion (0 to 3), and ascites (0 to 3), with higher scores indicating a worse condition on all scales

CONTACTS AND LOCATIONS:
Overall Officials: Dalia A Gomaa, MSc in clinical pharmacy, Principal Investigator — Tanta University
Locations (1):
- Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No